CLINICAL TRIAL: NCT06396390
Title: The Comparative Results of Progestin Primed Ovarian Stimulation (PPOS) and GnRH Antagonist Ovarian Stimulation Methods on IVF Outcomes
Brief Title: Comparison of Progestin Primed Ovarian Stimulation (PPOS) vs.GnRH Antagonist Methods on IVF Outcomes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nesta Clinic (Network)
Responsible Party: Principal Investigator, Emre Kar, Principal Investigator, Nesta Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024001
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: IVF; Fertility Issues; Infertility
Keywords: GnRH Antagonist; Progestin Primed Ovarian Stimulation; Infertility; Ovarian Stimulation
MeSH Terms: conditions — Infertility | interventions — Progestins; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progestin Primed Ovarian Stimulation (PPOS) (Experimental): In this patient group, progestin based protocol is going to be the main course of treatment.
  Interventions: Drug: Progestin
- GnRH Antagonist Stimulation (Active Comparator): In this patient group, GnRH Antagonist treatment protocol is going to be the main course of treatment.
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: Progestin — In this regimen, Dydrogesterone (Duphaston©; 10mg; Deva Holding, Tekirdag/Turkiye) 3x1 PO will be started on day 2 of menstrual cycle and will be continued until the trigger day. The patient's dosage will be tailored based on their BMI, AMH value, and the number of follicles observed during the ultrasound examination on the 2nd day of the menstrual cycle. For triggering, Choriogonadotropin-α (Ovitrelle©, 250 mcg/0.5 mL, Merck Serono S.p.A., Bari/Italy) 1 amp SC + Triptorelin Acetate (Gonapeptyl©, 0.1mg/mL, Ferring GmbH, Kiel/Germany) 2 amp SC will be used. All oocytes picked-up will be frozen.
  Other Names: Progestin Primed Ovarian Stimulation Protocol
  Arms: Progestin Primed Ovarian Stimulation (PPOS)
Drug: GnRH antagonist — In this regimen, Cetrorelix (Cetrotide©, 250 mcg/mL, Pierre Fabre Medicament Production, Idron, France) 1x1 SC will be started on day 7 of menstrual cycle and will be continued until the trigger day. For triggering, Choriogonadotropin-α (Ovitrelle©, 250 mcg/0.5 mL, Merck Serono S.p.A., Bari/Italy) 1 amp SC + Triptorelin Acetate (Gonapeptyl©, 0.1mg/mL, Ferring GmbH, Kiel/Germany) 2 amp SC will be used. All oocytes picked-up will be frozen.
  Other Names: GnRH Antagonist Ovarian Stimulation Protocol
  Arms: GnRH Antagonist Stimulation

SUMMARY:
The goal of this randomized clinical trial is to compare the effects of two different ovarian stimulation methods: Progestin Primed Ovarian Stimulation (PPOS) vs. GnRH Antagonist in embryologic outcomes of IVF Patients.

DETAILED DESCRIPTION:
The goal of this randomized clinical trial is to compare the effects of two different ovarian stimulation methods: Progestin Primed Ovarian Stimulation (PPOS) vs. GnRH Antagonist in embryologic outcomes of IVF Patients.

Ovarian stimulation will be conducted according to the assigned arm protocol.

Both artificially prepared and modified natural cycles will be eligible to be included and the choice will be done according to the doctor's preference and the patient's menstrual cycle regularity.

* For artificially prepared transfers, Estradiol Hemihydrate (Estrofem©, 2mg, Novo Nordisk, Malov/Denmark) 3x1 PO will be started on the day 2 of the menstrual cycle. After 12-14 days of usage, in order not to cancel the cycle, endometrial thickness needs measured at least 7mm and serum progesterone level < 1.5 ng/mL.
* For luteal support in addition to Progesterone (Progestan Dex©, 25mg, Kocak Farma İlaç ve Kimya Sanayi A.Ş., Istanbul, Turkiye) 2x1 SC once, with a 12-hour interval at day 14 of the menstrual cycle; Progesterone (Progestan©, 200mg, Kocak Farma İlaç ve Kimya Sanayi A.Ş., Istanbul, Turkiye) 2x1 PV will be started and continued for 5 days. Embryo transfer will be performed at 6th day. Estradiol Hemihydrate will be stopped on week 2 and progesterone support will be continued until the 8th week of gestation.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18 kg/m2 ve <35 kg/m2
* Couples that accept being included in the study
* Couple accepting thawed embryo transfer

Exclusion Criteria:

* Known chromosomal abnormality in either member of the couple
* Couples with unexplained infertility
* BMI > 30 kg/m2
* Mullerian malformations
* Undergoing oocyte cryopreservation for medical reasons (such as malignancies)
* Couple insists on fresh embryo transfer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Blastulation Rate | Day 5 or 6 after fertilization
  number of blastocysts up to day 6 / the number of fertilized 2PN embryos

SECONDARY OUTCOMES:
PGT Results | 14 days after blastocyte culture sampling
  Euploidy and aneuploidy rates
Ongoing pregnancy | on gestational week 12
  Fetal heart rate examination via USG
Live Birth Rate | 9 months
  For pregnancies resulted within the study period, live birth/embryo transfer count
Chemical Pregnancy | on day 11 after transfer
  Serum ß-hcg level

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bastu, M.D., Study Director — Owner
Locations (1):
- Nesta Clinic, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request for at least 2 years after publication.
Time Frame: At least 2 years after publication
Access Criteria: Upon request